CLINICAL TRIAL: NCT03719950
Title: Monocentric Study on the Quality of Life Among Adolescents With Attention Deficit/Hyperactivity Disorder
Brief Title: Study on the Quality of Life Among Adolescents With Attention Deficit/Hyperactivity Disorder
Acronym: QuaVAT
Status: Completed | Type: Observational
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH 2018-01; ID RCB 2018-A02303-52 (Other: ANSM (French competent authority))
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2020-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) with a overall prevalence of 5.3% is one of the most common neurobehavioral disorders in children. In the foreign literature, many studies bring to light in children and adolescents the negative impact of ADHD on overall quality of life. Some of these studies were able to identify the fact that the higher the age of ADHD children or adolescents, the lower the quality of life. Currently, to our knowledge, only a few European studies have demonstrated the negative impact of ADHD on the quality of life of children and adolescents. In addition, these studies used only questionnaires intended for parents and not for children or adolescents.

During a regular follow-up consultation with their referent child psychiatrist, adolescents accompanied by at least one of their parents will be informed of the modalities of our study. A newsletter will be delivered to parents and one to the adolescent. If neither the adolescent nor the parents is opposed to participate, the child psychiatrist will register the patient on the list of study participants. He will also fill out a medico-social information sheet about the adolescent as to summarize the data in the medical record. At the end of this consultation, in the waiting room, adolescents will answer questionnaires KIDSCREEN-27 and MSPSS; their parents will complete the CBCL questionnaire. These questionnaires will be handed to the secretary who will put them back in the patient's record. The KIDSCREEN-27, MSPSS and CBCL questionnaires as well as the medico-social information sheet will be source documents. The principal investigator or one of the associates investigators will complete the case report form from these source documents. For this purpose the data will be entered anonymously into a data entry software on a computer server secured by the Centre Psychothérapique de Nancy (CPN). Then, anonymous data from the software will be forwarded to Dr. Epstein of the Clinical Investigation Center for statistical analysis. The study will begin when the favourable opinion of the Ethical Research Comittees will be obtained and the study will last one year.

DETAILED DESCRIPTION:
Cross-sectional, descriptive epidemiological study based on single-centre trials

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 18 years
* Diagnosis of ADHD (f 90.0) ascertained by a child psychiatry according to CIM-10 criteria
* Seen by a child psychiatrist in consultation and accompanied by at least one of their parents
* Adolescents and at least one parent who has received enlightened information about the study
* Non-opposition to participate in the study gathered from at least one of their parents
* Patient affiliated or beneficiary of a social security scheme

Exclusion Criteria:

* Illiteracy of the parents or the adolescents
* Difficulties to understand french for the parents or the adolescents

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents (12 to 18 years old) with diagnosis of ADHD followed during regional child psychiatric consultation at Child department of Nancy University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The KIDSCREEN-27 | Day 0 (=day of inclusion = the only visit of the study)
  A shorter version of KIDSCREEN-52 which is Health-Related Quality of Life Questionnaire for Children and Adolescents aged from 8 to 18 years The adolescent will consult his child psychiatrist and after he will answer to the questionnaire KIDSCREEN-27 during estimated time of fifteen minutes.

SECONDARY OUTCOMES:
The Child Behavior Check List (CBCL) | Day 0 (=day of inclusion = the only visit of the study)
  The Child Behavior Check List assess behavioral or emotional psychopathological traits of children and adolescents aged 4 to 18 years. It composed of 118 items. The adolescent will consult his child psychiatrist and the parents will complete the Child Behavior Check List during about twenty minutes
The Multidimensional Scale of Perceived Social Support (MSPSS) | Day 0 (=day of inclusion = the only visit of the study)
  The MSPSS is a self-administered questionnaire designed to measure perceived social support. Composed of 12 items, the MSPSS measures perceived social support from three sources: family, friends and significant others. The adolescent will consult his child psychiatrist and after he will answer the MSPSS during about five minutes

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa WOLFF, Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Consultation régionale de pédopsychiatrie / Centre Psychothérapique de Nancy, Vandœuvre-lès-Nancy, Meurthe Et Moselle, France

IPD SHARING:
Plan to Share IPD: No